CLINICAL TRIAL: NCT06035406
Title: Pharmacokinetics and Safety of SP2086 in Subjects With Mild and Moderate Liver Impairment and Normal Liver Function.
Brief Title: A Trial of SP2086 With Hepatic Insufficiency
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP2086-117
Record Dates: First submitted 2023-09-07; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A: Retagliptin Phosphate Tablet (Experimental)
  Interventions: Drug: Retagliptin Phosphate Tablet
- Treatment group B: Retagliptin Phosphate Tablet (Experimental)
  Interventions: Drug: Retagliptin Phosphate Tablet
- Treatment group C: Retagliptin Phosphate Tablet (Experimental)
  Interventions: Drug: Retagliptin Phosphate Tablet

INTERVENTIONS:
Drug: Retagliptin Phosphate Tablet — Retagliptin Phosphate Tablet;100mg

SUMMARY:
This study used a single-dose, open design to compare the pharmacokinetics of subjects with mild and moderate liver impairment and subjects with normal liver function.

ELIGIBILITY:
Inclusion Criteria:

1. Sign informed consent before the test, and fully understand the test content, process and possible adverse reactions; And be able to complete the research according to the requirements of the test plan;
2. The subjects (including their partners) are willing to voluntarily take effective contraceptive measures from screening until 2 weeks after the last study drug administration, as specified in Appendix 1;
3. Age 18-70 years old (including the critical value), both male and female;
4. The weight of male subjects is not less than 50 kg, and the weight of female subjects is not less than 45 kg. Body mass index (BMI) : 18-32 kg/m2 (including the cut-off value);
5. (Only for subjects with normal liver function) The demographic mean of subjects in the normal liver function group (Group C) at screening must meet the following matching criteria:

   1. The body weight was matched with that of the liver function impairment group (group A + group B), with an average of ±10 kg;
   2. Age matching was performed with the liver function impairment group (group A + group B), and the mean was ±10 years old;
   3. Gender matching was performed with the liver function impairment group (group A + group B), with an average of ±1 cases;
6. (Only for subjects with normal liver function) Normal or abnormal clinical laboratory tests (blood routine, blood biochemistry, urine routine, coagulation function) have no clinical significance.
7. (Only for subjects with normal liver function) No prior serious primary diseases of major organs, including but not limited to gastrointestinal, respiratory, kidney, liver, nervous, blood, endocrine, tumor, immune, psychiatric or cardiovascular and cerebrovascular diseases
8. (Only for subjects with liver function impairment) Those who had not taken medication within 4 weeks prior to screening, or who had at least 4 weeks of stable medication for liver impairment and/or other comorbidification requiring long-term treatment
9. (Only for subjects with liver function impairment) Patients with liver insufficiency due to previous primary liver disease with Child-Pugh grade A or B.

Exclusion Criteria:

1. allergy, or known or suspected allergy to any of the ingredients in the investigational drug;
2. Smoking an average of more than 10 cigarettes per day in the 3 months before screening;
3. Alcoholics in the preceding 3 months, i.e. drinking more than 14 units of alcohol per week (1 unit = 285 mL for beer, 25 mL for spirits, or 100 ml for wine);
4. Drug abusers or drug urine screening test positive;
5. Blood donation or blood loss ≥400 mL within 3 months before screening, or receiving blood transfusion;
6. Major surgery or surgical incision not fully healed within 6 months prior to screening;
7. Had been exposed to DPP-IV inhibitors such as sitagliptin, saxagliptin, ligagliptin, vigagliptin within 1 month prior to administration;
8. Chinese herbal medicine was taken within 2 weeks before administration;
9. Have malignant tumors, or a history of malignant tumors within 5 years prior to screening (except for treated non-melanoma skin tumors with no signs of recurrence, and resected cervical intraepithelial neoplasia);
10. Patients with a history of severe hypoglycemia;
11. History of recurrent urinary tract infections or/and genital fungal infections;
12. Those who are expected to have a tendency to undergo surgery or be hospitalized during the trial;
13. Systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg at the time of screening;
14. 14.12- Patients with clinically significant ECG abnormalities (such as tachycardia/bradycardia requiring medical treatment, degree II-III atrioventricular block, or QTcF (male) ≥470ms, QTcF (female) ≥480ms), or other clinically significant abnormalities determined by the investigator and judged by the investigator to be unsuitable for participation in this study;
15. Female subjects were breastfeeding or had positive pregnancy results during the screening period or during the test;
16. 16. Serum creatinine values were estimated glomerular filtration rate calculated using the chronic kidney disease epidemiology collaboration CKD-EPI formula filtration rate eGFR) < 90 ml/min;
17. 17. Anyone who has consumed any food or drink containing alcohol (or positive breath test for alcohol), grapefruit juice/grapefruit juice, methylxanthine (such as coffee, tea, cola, chocolate, energy drinks), strenuous exercise or other factors affecting drug absorption, distribution, metabolism, excretion or other factors within 2 days prior to administration;
18. 18 Those who had any factors deemed inappropriate by the investigator to participate in the study.
19. (Only for subjects with normal liver function) Participants who have participated in clinical trials of any drug or medical device within 3 months prior to screening (subject to acceptance of the drug)
20. (Only for subjects with normal liver function) Hepatitis B surface antigen, hepatitis C virus antibody, human immunodeficiency virus antibody or syphilis antibody detection of any index screening positive excluded.
21. (Only for subjects with liver function impairment) Participants who have participated in clinical trials of any drug or medical device within 1 month prior to screening (subject to acceptance of the drug)
22. (Only for subjects with liver function impairment) A history of liver transplantation
23. (Only for subjects with liver function impairment) Subjects with liver failure, or liver cirrhosis with complications such as hepatic encephalopathy, hepatocellular carcinoma, esophageal variceal hemorrhage and other complications deemed inappropriate by the researchers to participate in the study
24. (Only for subjects with liver function impairment) In addition to the primary liver disease itself, a history of any serious disease, or a medical history or abnormalities that the investigator believes may affect the results of the trial, and/or clinically significant clinical laboratory tests, including, but not limited to, a history of circulatory, endocrine, nervous, digestive, urinary, or blood, immune, psychiatric, and metabolic disorders.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
PK parameters：Cmax； | 0hour to 72hours after the last dosing
PK parameters：AUC0-t； | 0hour to 72hours after the last dosing
PK parameters：AUC0-∞； | 0hour to 72hours after the last dosing

SECONDARY OUTCOMES:
PK parameters：Tmax； | 0hour to 72hours after the last dosing
PK parameters：t1/2； | 0hour to 72hours after the last dosing
PK parameters：CL/F； | 0hour to 72hours after the last dosing
PK parameters：V/F； | 0hour to 72hours after the last dosing
Incidence and severity of adverse events (AEs) | from screening to 168 hours after the last dosing

IPD SHARING:
Plan to Share IPD: Undecided